CLINICAL TRIAL: NCT02227888
Title: A Phase 1, Open-Label Study Evaluating the Pharmacokinetics of N91115 in Cystic Fibrosis Patients
Brief Title: PK Study of N91115 in Cystic Fibrosis Patients
Acronym: SNO3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nivalis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N91115-1PK-02
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Cystic Fibrosis
Keywords: CF; F508Del; Cavosonstat; N91115
MeSH Terms: conditions — Cystic Fibrosis | interventions — cavosonstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- N91115 (Experimental): Every 12 hour oral dosing of 50 mg N91115 for 14 days
  Interventions: Drug: N91115

INTERVENTIONS:
Drug: N91115 — S nitrosoglutathione reductase inhibitor
  Other Names: Cavosonstat

SUMMARY:
This Phase 1 study in F508del-CFTR homozygous CF patients is being conducted to assess the pharmacokinetics and absorption dynamics of N91115 compared with healthy subjects in order to identify an initial starting dose for Phase 2 trials.

DETAILED DESCRIPTION:
This is an open-label pharmacokinetic (PK) study of twice daily doses of 50 mg of N91115 administered for 14 days in F508del-CFTR homozygous CF patients. Six patients are planned for enrollment. Each patient will undergo screening (Day 28 to Day 3) and, if eligible, will return to the clinical site on Day 1 or optionally on Day 1. Eligibility will be reconfirmed and the patient will be admitted to a clinical research unit (CRU). Patients will stay overnight from Day 1 to Day 2 and will be discharged on Day 2 after all procedures and assessments are completed. Patients will return to the CRU as outpatients on Days 4, 7, 11, 14, and 15 for PK sample collection and other assessments. They will receive an oral dose of investigational medicinal product (IMP), N91115, twice daily on Days 1 through 14 and will be followed for PK through Day 15. Telephone calls to assess safety and ensure compliance with dosing will be made on days that patients do not make clinic visits (Days 3, 5, 6, 8, 9, 10, 12, and 13). Follow-up safety calls will then be made on Day 21 (adverse events) and Day 28 (serious adverse events only). Participation of an individual patient may last approximately 56 days from the time of screening until the end-of-study (Day 28) follow-up call.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of CF, homozygous for the F508del-CFTR mutation
2. Weight ≥ 40 kg at screening
3. FEV1 ≥ 40% of predicted normal for age, gender, and height (Hankinson standards) pre or post-bronchodilator value, at screening
4. Hematology, clinical chemistry, and urinalysis results with no clinically significant abnormalities that would interfere with the study assessments at screening

Exclusion Criteria:

1. History of any illness or condition that in the opinion of the investigator could confound the results of the study or pose additional risk when administered IMP
2. Any acute infection, including acute upper or lower respiratory infections and pulmonary exacerbations that require treatment or hospitalizations within 4 weeks of Study Day 1
3. Any change in chronic therapies for CF lung disease (e.g., Ibuprofen, Pulmozyme®, hypertonic saline, Azithromycin, TOBI®, Cayston®) within 4 weeks of Study Day 1
4. History, including the screening assessment, of ventricular tachycardia or ventricular arrhythmias
5. History, including the screening assessment, of prolonged QT and/or QTcF (Fridericia's correction) interval (> 450 msec)
6. History of solid organ or hematological transplantation
7. History of alcohol abuse or drug addiction (including cannabis, cocaine, and opioids) in the year prior to screening
8. Use of continuous (24 hr/day) or nocturnal supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 14 Days
  To assess the pharmacokinetics of N91115 after twice daily (q 12 h) doses given for 14 days by measuring plasma and urine concentrations of N91115 and its primary metabolite.

SECONDARY OUTCOMES:
Safety of dosing twice per day over 14 days | 14 Days
  To assess the safety of 14 twice daily (q 12 h) doses of N91115 in F508del-CFTR homozygous CF patients by monitoring, 12 lead ECG, Adverse events, Clinical safety laboratory tests (hematology, clinical chemistry, and urinalysis), Concomitant medications, Abbreviated physical examinations, Hemoglobin oxygen saturation (O2 Sat) by pulse oximetry, Spirometry, Telemetry, Vital signs, Weight

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shoemaker, MD, Study Director — Nivalis Therapeutics, Inc.
Locations (3):
- United States (3):
  - University of Alabama @ Birmingham, Birmingham, Alabama
  - Children's CO, Aurora, Colorado
  - National Jewish Health, Denver, Colorado